CLINICAL TRIAL: NCT01128998
Title: An Open-Label Phase I Dose-Escalation Study of Sorafenib Plus S-1 in Advanced Solid Tumors
Brief Title: Sorafenib Plus S-1 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICR-CT2008-01
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2012-08

CONDITIONS: Advanced Solid Tumors
Keywords: Sorafenib; S1; Advanced Solid Tumors; RD; MTD; DLT; PK; PG; Biomarker
MeSH Terms: interventions — Sorafenib; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1 and Sorafenib (Experimental)
  Interventions: Drug: Sorafenib; Drug: S-1

INTERVENTIONS:
Drug: Sorafenib — 1. Name: Sorafenib
  2. Dosage form: 200 mg / Tablet
  3. Dosing schedule: 200 mg bid, po, everyday, since Day 8 of Cycle 1
  Other Names: Nexavar
Drug: S-1 — 1. Name:S-1
  2. Dosage form: 20 mg or 25 mg / Capsule
  3. Dosing schedule: 20-40 mg/m2 bid,po, 14 days on & 7 days off
  Other Names: TS-1

SUMMARY:
Primary Objective:

1. To define the recommended dose for phase II study of S-1 combined with sorafenib
2. To evaluate the dose-limiting toxicities of the combination therapy

Secondary Objectives:

1. To characterize the pharmacokinetics (PK) of sorafenib and S-1 in the combination therapy
2. To investigate the impact of genetic polymorphisms of metabolic genes on the PK of sorafenib and S-1, respectively, as well as on the toxicity profile of the combination.
3. To determine the changes of biomarkers between pre- and post-treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven metastatic or locally advanced malignant solid tumors, which are refractory to current standard systemic treatment.
* Have measurable lesion.
* 20-75 y/o.
* ECOG performance score no more than 2.
* Life expectancy > 12 weeks.
* Adequate hematopoietic, hepatic and renal functions.

  1. Hemoglobin > 9.0 g/dl
  2. Absolute neutrophil count > 1,500/mm3
  3. Platelet count 100,000/ mm3
  4. Total bilirubin < 1.5 times the upper limit of normal (ULN)
  5. ALT and AST < 2.5 x ULN
  6. Serum creatinine < 1.0 x ULN
* Recovery from prior therapy that given > 4 weeks before enrolment.
* No pregnancy and breast-feeding.
* Signed informed consent.

Exclusion Criteria:

* Severe cardiovascular disorders.
* Pulmonary fibrosis or interstitial pneumonia.
* HIV infection.
* Active infection.
* Major anti-cancer treatment within 4 weeks of study entry.
* Exposure to the current investigational agent before.
* Known or suspected allergy to the current investigational agent.
* Unable to swallow oral medications.
* Substance abuse, medical, psychological or social conditions interfering with the patient's participation or evaluation of the study results.
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.
* Symptoms of bowel obstruction, malnutrition, splenomegaly.
* Receiving active anti-coagulant therapy.
* Patients with concurrent CYP 2A6 and/or CYP 3A4 or 3A5 inducers or inhibitors; a minimal of 2 weeks wash-out period required.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determination of MTD/RD | First two cycles

SECONDARY OUTCOMES:
Dose-limiting Toxicity | First two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D., Ph.D., Study Chair — National Institute of Cancer Research, National Health Research Institution, Taiwan
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan